CLINICAL TRIAL: NCT03179709
Title: Provider Perceptions of Neuromuscular Blockade in ARDS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeremy Kahn, Professor of Critical Care Medicine, University of Pittsburgh
Other Study IDs: 170115; U01HL123020 (NIH)
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Neuromuscular Blockade; Acute Respiratory Distress Syndrome
Keywords: Acute Respiratory Distress Syndrome; Neuromuscular Blockade; Interviews; Implementation Science
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intervention: The investigators will interview physicians, nurses, respiratory therapists and other clinicians who have cared for patients enrolled in the active treatment arm of ROSE.
  Interventions: Behavioral: Interview
- Control: The investigators will interview physicians, nurses, respiratory therapists and other clinicians who have cared for patients enrolled in the control treatment arm of ROSE.
  Interventions: Behavioral: Interview
- Refusal: The investigators will interview physicians who have refused to allow their patients to be enrolled in ROSE.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — The investigators will perform and analyze semi-structured interviews with enrolled participants.

SUMMARY:
The proposed study will use qualitative methodology to understand health care provider perceptions of neuromuscular blockade (NMB) in patients with Acute Respiratory Distress Syndrome (ARDS). To achieve this goal the investigators will conduct a prospective ancillary study at four clinical centers participating in the NHLBI PETAL network as part of the ROSE (Reevaluation of Systemic Early Neuromuscular Blockade) clinical trial (NCT02509078). Using thematic content analysis of semistructured interviews with health care providers caring for patients enrolled in the ROSE trial the investigators will determine the barriers to NMB use and develop a framework for future NMB adoption in ARDS.

DETAILED DESCRIPTION:
Efficient translation of clinical trial results into practice is an enduring challenge in critical care, with many critically ill patients not receiving evidence-based therapies proven to save lives. One approach to speed the translation of clinical trial evidence into practice is through qualitative research to better understand the barriers to evidence-based care and help design innovative interventions to overcome those barriers.. This work need not wait until the clinical trial is complete-an emerging literature highlights the value of qualitative research concurrent with the conduct of a clinical trial. Such research has several potential benefits, including facilitating implementation of the intervention in the real world, identifying the potential mechanism of action, and identifying contextual factors necessary for the treatments effectiveness.

The Reevaluation Of Systemic Early Neuromuscular Blockade (ROSE) study, conducted by the NHLBI PETAL Clinical Trials Network, is an ideal trial for which to perform a concurrent qualitative implementation study (NCT02509078). NMB has the potential to substantially reduce mortality in ARDS. Yet NMB remains incompletely adopted for reasons that are poorly understood but likely relate to clinical equipoise, historical concerns about safety, and the inherent difficulties in providing complex practices in the intensive care unit (ICU). A better understanding of provider views regarding NMB will provide essential data to aid interpretation of study results and design an implementation study should ROSE demonstrate a survival benefit with NMB.

To examine this issue the investigators will perform a prospective qualitative study using semi-structured interviews health care professionals providing direct care for patients enrolled in ROSE. A trained research coordinator will perform semi-structured interviews with consenting participants. Interviews will be transcribed and uploaded into commercially available qualitative data software. Trained qualitative researchers will read and code each interview based on Consolidated Framework for Implementation Research, a widely accepted conceptual theory of evidence-uptake.

ELIGIBILITY:
Inclusion Criteria:

* physician, nurse, respiratory therapist or clinical pharmacist providing direct care for patients enrolled in the ROSE study; or physician who refused entry of their patient into the ROSE study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Health care professionals with direct experience in either caring for patients enrolled in the ROSE trial (NCT02509078) or caring for patients with ARDS eligible for ROSe but not enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-18 (Actual); Study Completion 2018-03-18 (Actual)

PRIMARY OUTCOMES:
Barriers to adoption of NMB | 1 month post enrollment
  As a qualitative study, this study has no quantitative outcome measures. Provider perceptions of the knowledge, attitude, and behavioral barriers to adoption of early NMB in ARDS will be assessed using a semi-structured interview guide.
Contextual factors that influence the effectiveness of NMB | 1 month post enrollment
  As a qualitative study, this study has no quantitative outcome measures. Provider perceptions of the clinical and organizational factors that influence the impact of NMB on patient centered outcomes will be assessed using a semi-structured interview guide.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Kahn, MD, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No